CLINICAL TRIAL: NCT00127790
Title: CBT for Co-Morbid Insomnia and Chronic Pain: Sleep, Pain and Immune Function Outcomes
Brief Title: Treatment of Insomnia Secondary to Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Wilfred Pigeon, Asst Prof, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160743209; F32NS049789 (NIH); K23NR010408 (NIH); R21AG023956; R24AG031089 (Other: Rochester Center for MindBody Research); R21AG023956 (NIH)
Record Dates: First submitted 2005-08-03; First posted 2005-08-08 (Estimated); Results first posted 2012-10-17 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-09

CONDITIONS: Insomnia; Pain
Keywords: Insomnia; Sleep; Pain; Pain, Chronic; Behavior Therapy; CBT; CBT-I; cognitive-behavioral
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Pain; Chronic Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CBT for Insomnia (CBT-I) (Active Comparator): Cognitive-Behavioral Therapy for Insomnia (CBT-I)consisting of 10 individual sessions and including sleep education, sleep restriction therapy, stimulus control therapy, sleep hygiene, cognitive therapy, relaxation training and relapse prevention.
  Interventions: Behavioral: CBT for Insomnia (CBT-I)
- CBT for Pain (CBT-P) (Active Comparator): Cognitive-Behavioral Therapy for Pain (CBT-P)consisting of 10 individual sessions and including pain education, pacing strategies, problem solving, goal setting, cognitive therapy, relaxation training and relapse prevention.
  Interventions: Behavioral: CBT for Pain (CBT-P)
- CBT for Insomnia & Pain (CBT-I/P) (Experimental): Combined Cognitive-Behavioral Therapy for Insomnia & Cognitive-Behavioral Therapy for Pain (CBT-I/P)over 10 individual sessions.
  Interventions: Behavioral: CBT for Insomnia (CBT-I); Behavioral: CBT for Pain (CBT-P)
- Wait-List Control (WL) (No Intervention): Waitlist Control condition (WL) with no contact during the intervention period.

INTERVENTIONS:
Behavioral: CBT for Insomnia (CBT-I)
  Other Names: Cognitive-Behavioral Therapy for Insomnia (CBT-I)
  Arms: CBT for Insomnia & Pain (CBT-I/P); CBT for Insomnia (CBT-I)
Behavioral: CBT for Pain (CBT-P)
  Other Names: Cognitive-Behavioral Therapy for Pain (CBT-P)
  Arms: CBT for Insomnia & Pain (CBT-I/P); CBT for Pain (CBT-P)

SUMMARY:
Several studies have shown that behavioral therapy for chronic pain can be beneficial for chronic pain and that behavioral therapy for insomnia can be beneficial for insomnia. However, seldom do chronic pain patients with insomnia receive a behavioral treatment for insomnia. The purpose of this study is to evaluate whether treatment for insomnia is helpful for pain and whether treatment for pain is helpful for insomnia. It will also assess whether a combined treatment is any more or less effective for pain or for sleep. Finally, the study will assess whether any of these treatments leads to improvements in immune function.

DETAILED DESCRIPTION:
The investigators' primary goal is to assess the extent to which three forms of cognitive-behavioral treatment (CBT for insomnia, CBT for pain, and combined insomnia & pain) diminishes insomnia symptoms in patients with chronic pain compared to a group not receiving CBT. This will be evaluated in a randomized trial with before and after evaluations using standard sleep diary measures of sleep continuity.

The investigators' secondary goal is to assess whether treatment responses to any of the interventions are associated with alterations in immune function.

The investigators' tertiary goals are to evaluate whether improved sleep has effects on patient reports of pain severity, frequency, and tolerability as well as on mood and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Ages 35-75
* Chronic non-malignant painful condition of the spine of > 6 months duration
* Insomnia (> 30 minutes sleep latency and/or wake after sleep onset time for > 3 days/week for > 6 months)
* Insomnia developed after the onset of the painful condition
* Preferred sleep phase between 10:00 p.m. and 8:00 am
* On stable medical regimen for medical and pain conditions (no surgery planned)
* Willingness to discontinue hypnotic medications

Exclusion Criteria:

* Unstable medical or psychiatric illness
* History of seizures
* Evidence of active illicit substance use or fitting criteria for ethanol (ETOH) abuse or dependence
* Symptoms suggestive of sleep disorders other than insomnia
* Polysomnographic data indicating sleep disorders other than insomnia
* Inadequate language comprehension
* Fibromyalgia
* Pregnancy

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-06; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilfred R. Pigeon, Ph.D, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Sleep Research Laboratory, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men and women aged 35-75 experiencing chronic pain and insomnia were recruited from the community through newspaper advertisements and from local pain clinics via recruitment flyers.
Pre-assignment Details: Participants completed intake interview, physical exam, clinical chemistries and toxicology screens; completed daily pain-sleep diaries for two weeks; and then underwent polysomnography. Seven subjects were excluded prior to randomization (4 due to sleep apnea, 1 did not meet pain severity criteria, and 2 subsequently declined to participate).
Groups:
- Cognitive-Behavioral Therapy for Insomnia (CBT-I): Cognitive-Behavioral Therapy for Insomnia (CBT-I)consisting of 10 individual sessions and including sleep education, sleep restriction therapy, stimulus control therapy, sleep hygiene, cognitive therapy, relaxation training and relapse prevention.
- Cognitive-Behavioral Therapy for Pain (CBT-P): Cognitive-Behavioral Therapy for Pain (CBT-P)consisting of 10 individual sessions and including pain education, pacing strategies, problem solving, goal setting, cognitive therapy, relaxation training and relapse prevention.
- Cognitive-Behavioral Therapy for Insomnia & Pain (CBT-I/P): Cognitive-Behavioral Therapy for Insomnia & Pain (CBT-I/P)consisting of 10 individual sessions and including sleep education, pain education, sleep restriction therapy, stimulus control therapy, sleep hygiene, pacing strategies, problem solving, goal setting, cognitive therapy, relaxation training and relapse prevention.
Period: Pre-Treatment
Arm/Group | Cognitive-Behavioral Therapy for Insomnia (CBT-I) | Cognitive-Behavioral Therapy for Pain (CBT-P) | Cognitive-Behavioral Therapy for Insomnia & Pain (CBT-I/P) | Wait-List Control (WL)
Started | 6 (7 enrolled subjects were withdrawn prior to randomization; 21 of 28 enrolled were randomized.) | 5 | 6 | 4
Completed | 6 | 5 | 6 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Post-Treatment
Arm/Group | Cognitive-Behavioral Therapy for Insomnia (CBT-I) | Cognitive-Behavioral Therapy for Pain (CBT-P) | Cognitive-Behavioral Therapy for Insomnia & Pain (CBT-I/P) | Wait-List Control (WL)
Started | 6 | 5 | 6 | 4
Completed | 6 | 5 | 6 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive-Behavioral Therapy for Insomnia (CBT-I) | Cognitive-Behavioral Therapy for Pain (CBT-P) | Cognitive-Behavioral Therapy for Insomnia & Pain (CBT-I/P) | Wait-List Control (WL) | Total
Number analyzed (Participants) | 6 | 5 | 6 | 4 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 6 | 4 | 20
  >=65 years | 0 | 1 | 0 | 0 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 45.7 (8.2) | 55.8 (9.8) | 50.5 (8.5) | 52.3 (1.0) | 50.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6 | 2 | 14
  Male | 2 | 3 | 0 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 6 | 4 | 21

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity
Description: Total Score from the 7-item Insomnia Severity Index where total score ranges from 0-28 and higher scores indicate greater severity of insomnia.
Time Frame: Pre to Post Treatment Change (Over an average of approximately 10 weeks)
Population: completed the intervention and self report instruments
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive-Behavioral Therapy for Insomnia (CBT-I) | Cognitive-Behavioral Therapy for Pain (CBT-P) | Cognitive-Behavioral Therapy for Insomnia & Pain (CBT-I/P) | Wait-List Control (WL)
Number analyzed (Participants) | 6 | 5 | 6 | 4
units on a scale | 6.0 (1.9) | 12.8 (1.1) | 4.4 (1.0) | 13.0 (1.7)
Statistical Analysis 1: Comparison: Cognitive-Behavioral Therapy for Insomnia (CBT-I) vs Wait-List Control (WL); Two-tailed comparison of pre-post scores; Test type: Superiority or Other; p = 0.010, Generalized Estimating Equations; Mean Difference (Final Values) = 7.0
Statistical Analysis 2: Comparison: Cognitive-Behavioral Therapy for Pain (CBT-P) vs Wait-List Control (WL); Two-tailed comparison of pre-post scores; Test type: Superiority or Other; p = 0.581, Generalized Estimating Equations; Mean Difference (Final Values) = 0.5
Statistical Analysis 3: Comparison: Cognitive-Behavioral Therapy for Insomnia & Pain (CBT-I/P) vs Wait-List Control (WL); Two-tailed comparison of pre-post scores; Test type: Superiority or Other; p = 0.011, Generalized Estimating Equations; Mean Difference (Final Values) = 8.6

2. Primary Outcome: Pain Severity
Description: Multidimensional Pain Inventory - Pain Severity SubScale score. The subscale consists of 3 items with a total subscale score ranging from 0-18 with higher values indicating greater pain severity.
Time Frame: Pre to Post Treatment Change (Over an average of approximately 10 weeks)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive-Behavioral Therapy for Insomnia (CBT-I) | Cognitive-Behavioral Therapy for Pain (CBT-P) | Cognitive-Behavioral Therapy for Insomnia & Pain (CBT-I/P) | Wait-List Control (WL)
Number analyzed (Participants) | 6 | 5 | 6 | 4
units on a scale | 11.0 (2.3) | 6.2 (1.7) | 8.8 (1.9) | 7.5 (1.0)
Statistical Analysis 1: Comparison: Cognitive-Behavioral Therapy for Insomnia (CBT-I) vs Wait-List Control (WL); Two-tailed comparison of pre-post scores; Test type: Superiority or Other; p = 0.33, Generalized Estimating Equations; Mean Difference (Final Values) = 3.5
Statistical Analysis 2: Comparison: Cognitive-Behavioral Therapy for Pain (CBT-P) vs Wait-List Control (WL); Two-tailed comparison of pre-post scores; Test type: Superiority or Other; p = 0.112, Generalized Estimating Equations; Mean Difference (Final Values) = -1.2
Statistical Analysis 3: Comparison: Cognitive-Behavioral Therapy for Insomnia & Pain (CBT-I/P) vs Wait-List Control (WL); Two-tailed comparison of pre-post scores; Test type: Superiority or Other; p = 0.737, Generalized Estimating Equations; Mean Difference (Final Values) = 1.3

3. Primary Outcome: IL-6
Description: Circulating levels of Interleukin-6 (IL-6)from plasma drawn in the morning. Values are presented as picograms per milliliter (pg/mL) and can range from 0 to 500, though tend to be in the range of 0-10. Higher values indicate higher amounts of circulating levels of IL-6, a marker of increased inflammatory processes.
Time Frame: Pre to Post Treatment Change (Over an average of approximately 10 weeks)
Population: Subjects completing blood draws to obtain plasma. One subject in the CBT-I&P condition did not complete blood draws.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Cognitive-Behavioral Therapy for Insomnia (CBT-I) | Cognitive-Behavioral Therapy for Pain (CBT-P) | Cognitive-Behavioral Therapy for Insomnia & Pain (CBT-I/P) | Wait-List Control (WL)
Number analyzed (Participants) | 6 | 5 | 5 | 4
pg/mL | 0.7 (0.2) | 1.6 (1.0) | 1.2 (0.2) | 1.2 (0.3)
Statistical Analysis 1: Comparison: Cognitive-Behavioral Therapy for Insomnia (CBT-I) vs Wait-List Control (WL); Two-tailed comparison of pre-post scores; Test type: Superiority or Other; p = 0.063, Generalized Estimating Equations; Mean Difference (Final Values) = 0.5
Statistical Analysis 2: Comparison: Cognitive-Behavioral Therapy for Pain (CBT-P) vs Wait-List Control (WL); Two-tailed comparison of pre-post scores; Test type: Superiority or Other; p = 0.786, Generalized Estimating Equations; Mean Difference (Final Values) = 0.4
Statistical Analysis 3: Comparison: Cognitive-Behavioral Therapy for Insomnia & Pain (CBT-I/P) vs Wait-List Control (WL); Two-tailed comparison of pre-post scores; Test type: Superiority or Other; p = 0.039, Generalized Estimating Equations; Mean Difference (Final Values) = 0.0

4. Secondary Outcome: Depression Severity
Description: Total score from the 20-item Center for Epidemiologic Studies Depression Scale-revised where the total score ranges from 0-60 and higher scores indicate greater depression severity.
Time Frame: Pre to Post Treatment Chnage (Over an average of approximately 10 weeks)
Population: participants who completed intervention and pre and post treatment assessments
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive-Behavioral Therapy for Insomnia (CBT-I) | Cognitive-Behavioral Therapy for Pain (CBT-P) | Cognitive-Behavioral Therapy for Insomnia & Pain (CBT-I/P) | Wait-List Control (WL)
Number analyzed (Participants) | 6 | 5 | 5 | 4
units on a scale | 2.3 (1.9) | 10.2 (2.9) | 4.4 (1.8) | 17.6 (1.2)
Statistical Analysis 1: Comparison: Cognitive-Behavioral Therapy for Insomnia (CBT-I) vs Wait-List Control (WL); Two-tailed comparison of pre-post scores; Test type: Superiority or Other; p = 0.016, Generlaized Estimating Equations; Mean Difference (Final Values) = 15.2
Statistical Analysis 2: Comparison: Cognitive-Behavioral Therapy for Pain (CBT-P) vs Wait-List Control (WL); Two-tailed comparison of pre-post scores; Test type: Superiority or Other; p = 0.187, Generalized Estimating Equations; Mean Difference (Final Values) = 7.4
Statistical Analysis 3: Comparison: Cognitive-Behavioral Therapy for Insomnia & Pain (CBT-I/P) vs Wait-List Control (WL); Two-tailed comparison of pre-post scores; Test type: Superiority or Other; p = 0.015, Generalized Estimating Equations; Mean Difference (Final Values) = 13.2

ADVERSE EVENTS:
Arm/Group | Cognitive-Behavioral Therapy for Insomnia (CBT-I) | Cognitive-Behavioral Therapy for Pain (CBT-P) | Cognitive-Behavioral Therapy for Insomnia & Pain (CBT-I/P) | Wait-List Control (WL)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/6 | 0/4

LIMITATIONS AND CAVEATS:
The foremost limitation of this pilot study is its small sample size, particularly for a four-arm design. Accordingly, a cautious approach to the interpretation of the findings is warranted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No